CLINICAL TRIAL: NCT05668221
Title: Multidisciplinary Prehabilitation to Improve Frailty and Functional Capacity in High-risk Elective Surgical Patients: a Retrospective Pilot Study
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, WONG MAN KIN, Principal Investigator, Honorary Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2021.493-T
Record Dates: First submitted 2022-12-13; First posted 2022-12-29 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty | interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Prehabilitation — Prehabilitation includes exercise prescription, cognitive function assessment and training, nutritional optimisation at least 4 weeks prior to surgery

SUMMARY:
Frailty is a multidimensional syndrome in which multiple small physiological deficits accumulate gradually, resulting in a loss of physiological reserve and adaptability, putting a patient that is exposed to stressor at a higher risk of adverse outcomes. Both pre-frailty and frailty are associated with worse outcomes and higher healthcare costs. With the potential "teachable" moment from the long surgical waiting time in Hong Kong, the effect of a prehabilitation program incorporated into clinical care pathway in high-risk frail patients undergoing elective major surgery were evaluated.

DETAILED DESCRIPTION:
Traditionally in surgical practice, the decision to proceed to surgery is made between the surgeons and the patients. Whenever necessary, the patients are sent to other specialties (eg. anaesthesiologists, physicians, dietitians, physiotherapists) for consultation and optimization before elective surgery. This approach is acceptable for the majority of fit patients, it can however be unsatisfactory for high-risk frail patients undergoing major surgical procedures. Hong Kong is facing an aging population. According to the 2016-based population projections published by the Census and Statistics Department, the pace of population aging in Hong Kong will keep on ramping up in the coming 20 years or so. Between 2018 and 2038, the size and share of the elderly population will almost double from 1.27 million and 17.9% to 2.44 million and 31.9% respectively. With aging, there is an increase in frailty and a loss in functional and physiological reserve and adaptability, putting a patient that is exposed to a stressor, such as a major operation, at a higher risk of adverse outcomes. Frailty is associated with two to six- fold increased risk of major adverse cardiac and cerebrovascular events, longer stays in intensive care unit and hospital, a 1-year mortality. Pre-frail patients are also at risk of poor outcomes. Compared to non-frail patients, pre-frail patients (Clinical Frailty Score 4) had longer ICU stays, longer hospital stays, higher risk of postoperative stroke and a high risk of in-hospital mortality. Malnutrition and sedentary lifestyle are common in frail elderly patients. These have been demonstrated to be a recognizable risk factor of poor postoperative outcomes. It is therefore necessary to have a multidisciplinary team to manage frailty preoperatively.

Prehabilitation is a multidisciplinary and multimodal approach involving anaesthesiologists, physicians, physiotherapists, occupational therapists and dietitians that aims to optimize functional capacity, nutritional status and emotional resilience before surgery, so as to enable the patients to better withstand perioperative stress. It encompass individualized aerobic and resistance training to enhance cardiopulmonary fitness, dietary interventions to counteract the catabolic state of surgery, emotional support to improve resilience and advice on behavioural changes such as cessation of smoking and alcohol abuse. In the literature, prehabilitation has well been reported to enhance functional capacity before and after surgery. In particular, exercise training has been shown to improve various aspects of physical function of the frail elderly (eg. muscle strength, body composition, mobility, functional status and fall prevention). Tailored exercise training is therefore expected to improve physical fitness and increase functional capacity so that patients can better withstand the stress of surgery. In a systematic review, prehabilitation before orthopaedic surgery have beneficial effects in improving strength, flexibility, balance and speed in 5 out of 7 randomized controlled trials. Regarding postoperative clinical outcomes such as length of stay, readmission rate and postoperative complications rate, evidence demonstrated an association between physical fitness improvement and a lower rate and severity of complications. Despite the heterogenicity in study design and modalities of prehabilitation program, the positive effect of prehabilitation on perioperative functional fitness has been shown across a wide variety of surgical procedures, including abdominal aortic aneurysm repair, esophagectomy, cystectomy, liver resection and colorectal surgery. In general, individuals who have been frail and having a sedentary activity level would benefit the most from prehabilitation program. Preoperative malnutrition can be due to inadequate intake and high requirements from the disease process that results in reduced body mass, strength and function and a reduced ability to mount an immunological defense. All these can be significant in the high catabolic state perioperatively for the healing process and the systemic inflammatory response to surgery. Preoperative malnutrition is associated with many adverse outcomes. After adjusting for active smoking status, preoperative malnutrition was associated with postoperative complications after pneumonectomy and hepatectomy, a longer length of stay in hospital, higher readmissions within 28 days and a higher mortality up to 90 days after surgery. Nutritional prehabilitation therefore helps prepare and optimize the patients' nutritional status for surgery and recovery.

The timing and duration of prehabilitation program can affect the risk of postoperative outcomes. An ideal duration of prehabilitation has not been established and there is a large heterogenicity in duration from the literature. But in general, a minimum of three to four weeks is required to have an effect of physical fitness. Despite the need for novel resources, economic evaluation suggested that prehabilitation could be a cost-effective approach, the resulting benefits in short- and medium-term outcomes offset the costs of additional resources.

Most of the "fast-track" surgical pathways focus on intraoperative and postoperative measures to enhance recovery, and the traditional rehabilitation approach is to operate first and then intervene. However, postoperative pain, fatigue and wound care impede the efficiency of rehabilitation measures such as physiotherapy and nutritional program. Therefore, it would be more ideal to start intervention before surgery while patients can be more actively engaged in the process of perioperative care and functional improvement. The earlier the patients can be engaged, the greater the likelihood of having a meaningful impact and the less likely to affect the surgical schedule. The waiting time for surgery creates a window of opportunity to prepare the patients for prehabilitation by addressing problems of physical fitness, nutritional status and emotional distress. By re-engineering our preoperative assessment clinic and integration within the prehabilitation clinic, we are more able to risk stratify and identify high-risk patients at the time of preoperative evaluation. A common and one-stop platform can be shared by a multidisciplinary perioperative team with seamless communications, which reduces the chance of high-risk patients being bounced between independent consultations.

Changing the present structure and logistics of preoperative assessment clinic requires active participation of the stakeholders involved in perioperative care. Surgeons need to refer patients to anaesthesiologists as early as possible for further screening into prehabilitation program. Anaesthesiologists need to have new assessment strategies for functional capacity that are not traditionally used in routine preoperative assessment clinic. Physiotherapist, occupational therapist and dietitians should ideally set up a one-stop service model to minimize patient travel. Effective implementation requires buy-in from hospital administrators, investing resources to support this value-based approach. Therefore, the investigators will conduct a pilot retrospective observational study to evaluate the feasibility and impact of prehabilitation on our study participants before major elective surgery. In particular, for the feasibility part, the investigators aim to (1) estimate recruitment, attrition and adherence rate, and (2) ensure safety of prehabilitation. For the pilot part, the investigators aim to identify if there are any changes on the outcomes after the prehabilitation intervention, and (2) identify estimates of variance for sample size calculation for future randomized trials.

ELIGIBILITY:
Inclusion Criteria:

* Procedure-specific: major hepatectomy (resection of 3 or more Couimaud's segments), pancreaticoduodenectomy, esophagectomy and radical cystectomy
* Patient-specific: age 50 or above, undergoing elective major procedures, together with one of the followings:

  1. American Society of Anaesthesiologists physical status score >=3
  2. Pre-frail to moderately frail patients with a Clinical Frailty Scale 3-6 at the time of assessment at prehabilitation clinic
  3. 6-minute walk test distance <400 meters
  4. Duke Activity Status Index <34
  5. Malnutritional Screening Tool score >=2

Exclusion Criteria:

* Patients with unstable angina or unstable cardiac syndrome (New York Heart Association Class IV, critical left main coronary disease, hospitalization for arrhythmias, congestive heart failure or acute coronary syndrome before assessment at prehabilitiation clinic)
* Patients with left ventricular outflow obstruction (severe aortic stenosis, hypertrophic cardiomyopathy)
* Chronic obstructive pulmonary disease GOLD stage IV
* Abdominal aortic aneurysm >8.0cm or suspected dissecting or leaking aortic aneurysm
* Cognitive deficits unable to comply with study procedures, physical limitations that would prelude rehabilitation and inability to regularly attend prehabilitation sessions.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Local Hong Kong population, usually elderly frail patients with the above criteria, booked for elective major operation and seen at prehabilitation clinic at least 4 weeks prior to procedure
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Up to 1 year after the first case recruitment
  Number of patients successfully enrolled into prehabilitation program divided by the number of patients attending prehabilitation clinic
Attrition rate | Through study completion, an average of 18 months after the first recruitment
  Number of patients who dropped out divided by the number of patients enrolled into prehabilitation program
Adherence of patients to prehabilitation program | Through study completion, an average of 18 months after the first recruitment
  Number of patients completed prehabilitation program divided by the number of patients enrolled

SECONDARY OUTCOMES:
6-minute walk test distance | 1 year
  Distance in metre walked by the patient over 6 minute. The patient walks back and forth at a standardised 30 meter distance
Calculated peak oxygen uptake | 1 year
  Calculated from 6-minute walk test distance using standardised formula
Hand grip strength | 1 year
  Measurement using a hand-grip strength meter by physiotherapy. The strength is in the unit kilogram. Left and right hand grip strength will be measured separately
30 second chair stand test | 1 year
  Patient is asked to sit and stand from a chair as many times as possible within 30 second
Time-up-and-go test | 1 year
  Time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees
Depression Anxiety Stress Scale | 1 year
  A standardised questionnaire measuring the degree of depression, anxiety and stress. An assessment of emotional resilience. The scale score ranges from 0 to 126, including 42 items. The higher score corresponds to worse performance
Body mass index | 1 year
  A measure of nutritional status. Weight in kilogram and height in meter will be combined to report body mass index in kg/m^2
muscle mass | 1 year
  A measure of nutritional status
Percentage body fat | 1 year
  A measure of nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: Man Kin Wong, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data will be kept confidential in locked drawers within the principle investigator's office. It can only be assessed by the principle investigator

REFERENCES:
- [Derived] Wong HMK, Qi D, Ma BHM, Hou PY, Kwong CKW, Lee A; Prehab Study Group. Multidisciplinary prehabilitation to improve frailty and functional capacity in high-risk elective surgical patients: a retrospective pilot study. Perioper Med (Lond). 2024 Jan 23;13(1):6. doi: 10.1186/s13741-024-00359-x. PMID 38263053

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT05668221/Prot_SAP_000.pdf